CLINICAL TRIAL: NCT00307684
Title: An Open International Multicentre Long-Term Follow Up Study to Evaluate Safety of Prolonged Release OROS Methlyphenidate in Adults With Attention Deficit Hyperactivity Disorder
Brief Title: Open Label, Multicentre Extension Study of Protocol 42603ATT3002 to Evaluate Safety of Prolonged Release OROS Methlyphenidate in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR011068; NCT00980499 (obsolete NCT alias)
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; Adult; Long term safety; Efficacy; Quality of life
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Experimental): open label PR OROS methylphenidate Flexible dosage MPH (18 to 90 mg/day) for 72 weeks (108 weeks for Germany)
  Interventions: Drug: open label PR OROS methylphenidate
- 002 (Experimental): double blind PR OROS methylphenidate 18 36 54 72 or 90 mg/day once daily for 4 weeks
  Interventions: Drug: double blind PR OROS methylphenidate
- 003 (Placebo Comparator): double blind placebo matching placebo tablets once daily for 4 weeks
  Interventions: Drug: double blind placebo

INTERVENTIONS:
Drug: double blind placebo — matching placebo tablets once daily for 4 weeks
  Arms: 003
Drug: double blind PR OROS methylphenidate — 18, 36, 54,72 or 90 mg/day once daily for 4 weeks
  Arms: 002
Drug: open label PR OROS methylphenidate — Flexible dosage MPH (18 to 90 mg/day) for 72 weeks (108 weeks for Germany)
  Arms: 001

SUMMARY:
Trial 42603ATT3004 is an open-label extension study to clinical trial 42603ATT3002 (NCT00246220). In trial 42603ATT3002 the efficacy and safety of OROS methylphenidate was assessed in adult subjects with Attention Deficit Hyperactivity Disease (ADHD). ADHD is a developmental disorder beginning in childhood and characterized by developmentally inappropriate inattention, hyperactivity and impulsiveness. Data on the number of adult patients with ADHD is limited, but it is estimated that approximately 50% of children with ADHD will have symptoms also in adhulthood. The drug tested in this trial is OROS methylphenidate. The active ingredient is methylphenidate and the tablet is designed to release the active ingredient gradually to ensure an effect, which lasts up to 12 hours. Trial 42603ATT3002 consisted of a 5-week period, where subjects were assigned to either receive placebo (empty drug) or one out of three different dosages of OROS methylphenidate. This 5-week period was followed by a 7-week period, where patients received OROS methylphenidate at their optimal dose. In study 42603ATT3004, subjects who complete 42603ATT3002 are followed for a period of at least 52 weeks to evaluate safety and tolerability of OROS methylphenidate in patients who are treated with OROS methylphenidate over a long period of time.

Amendment: At the end of the open-label period of the present study 42603ATT3004, patients are enrolled into a double-blind placebo-controlled period, which lasts an additional 4 weeks. The purpose of this double-blind placebo-controlled period is to evaluate the maintenance of effect under continued treatment with OROS methlyphenidate in comparison to treatment cessation in those patients, who are randomized into the placebo-group.

DETAILED DESCRIPTION:
This is an open label, multicentre extension study to trial 42603ATT3002. Patients, who were enrolled to trial 42603ATT3002 must have had a diagnosis of ADHD with some symptoms already present at the age of 7 and continuing in adulthood. The patients must have had at least mild to moderate symptoms of ADHD. In trial 42603ATT3002 the efficacy and safety of three fixed dosages of the study drug OROS methlyphenidate (MPH) was compared with placebo in adult subjects with ADHD in a double-blind phase. This double-blind phase was followed by an open-label phase, which was designed to assess the safety and tolerabiltiy of the study drug OROS methylphenidate in these subjects, when they got a dose, which was optimal to control their symptoms. In trial 42603ATT3004 patients are enrolled who completed the open-label phase of trial 42603ATT3002. Trial 42603ATT3004 is designed to assess the long-term safety and tolerabilty of OROS methylphenidate over a period of 52 weeks at a dose, which is optimal to control the symptoms. Patients may enter the extension study 42603ATT3004 at Visit 8 (End-of-Phase Visit, Open Label) of the 42603ATT3002 study as long as the patient has given informed consent prior to the visit being performed. Visit 8 data may then serve as baseline data for the extension study. These patients should continue treatment at the same optimal dosage of PR OROS methylphenidate as was attained during the open label phase of protocol 42603ATT3002. Patients who complete the 42603ATT3002 study, including post-study visit, may enter the extensions study up to 30 calendar days from the last dosing of open label trial medication of the 42603ATT3002 study. Patients should be titrated accordingly to their optimal dose attained in study 42603ATT3002. Patients will be assessed at regular intervals for at least 52 weeks.

Amendment: At completion of the open-label phase, patients can participate in a double-blind placebo-controlled phase, provided that they are giving written informed consent. At inclusion to the double-blind placebo-controlled phase, patients are assigned to one of two treatment arms by chance. One treatment arm will continue taking the same treatment at the same daily dose as during the open-label period. The other treatment arm will receive placebo treatment. As placebo, an inactive formulation or an empty treatment will be used. During the double-blind placebo-controlled phase, patients are asked to return to their doctor's office every other week. During these visits, physical examinations will be made, efficacy measures will be taken by means of questionnaires, that need to be completed either by the treating physician or the patient and any unwanted side effect will be recorded and treated if needed. One week after the end of the double-blind, placebo-controlled phase, patients have to return one more time to their doctor's office for the so called post-study visit, during which an additional physical examination will be performed and additional safety and efficacy parameters will be assessed.Patients will be assessed at regular intervals for at least 52 weeks. Daily oral dosages of 18, 36, 54, 72 and 90mg will be available and may be increased or decreased by 18mg increments based on clinical observations of response and tolerability for at least 52 weeks. Amendment: During the double-blind, placebo-controlled phase, patients will receive either active treatment at the previously assessed optimal dose or placebo tablets for a total of 4 weeks. Both treatments (active or placebo) are taken by mouth once per day in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed study CR002479 (42603ATT3002), according to protocol
* Diagnosis of ADHD according to the Diagnostic and Statistical Manual of Mental Diseases, Fourth Edition (DSM-IV)1 and confirmed by the Conners' Adult ADHD Diagnostic Interview for DSM IV (CAADID)
* Healthy on the basis of physical examination, medical history
* Patient is able to comply with the study visit schedule and willing and able to complete the protocol-specified assessments
* Amendment (double-blind placebo-controlled period): written informed consent
* patient must have completed at least 52 weeks of open-label treatment and must have been on a stable daily dose of (PR) OROS methlyphenidate prior to inclusion to this phase

Exclusion Criteria:

* Patient is known to be a non-responder to methylphenidate, or patient has a child known to be a non-responder to methylphenidate
* Allergy or hypersensitivty to methlyphenidate
* Any clinically unstable psychiatric condition including but not limited to the following: acute mood disorder, bipolar disorder, acute obsessive-compulsive disorder (OCD), Anti-social personality disorder, borderline personality disorder
* Use of other anti-depressants (unless patient has been on a stable dosage during the 42603ATT3002 trial, in which case treatment may continue as long as dosage remains unchanged for the duration of the study) or mood stabilisers (e.g. anti-epileptics, lithium)
* Any medication likely to interfere with safe administration of methylphenidate, or any conditions that are contraindicated for use of methlyphenidate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (21):
- Paris, France
- Germany (11):
  - Ahrensburg
  - Aschaffenburg
  - Berlin
  - Cologne
  - Essen
  - Freiburg I. Br.
  - Homburg
  - Mannheim
  - Ottobrunn bei München
  - Saarbrücken
  - Würzburg
- Netherlands (2):
  - Nijmegen
  - The Hague
- Norway (2):
  - Drammen
  - Ottestad
- Portugal (2):
  - Cascais
  - Porto
- Barcelona, Spain
- Switzerland (2):
  - Basel Bs
  - Zurich

REFERENCES:
- [Derived] Boesen K, Paludan-Muller AS, Gotzsche PC, Jorgensen KJ. Extended-release methylphenidate for attention deficit hyperactivity disorder (ADHD) in adults. Cochrane Database Syst Rev. 2022 Feb 24;2(2):CD012857. doi: 10.1002/14651858.CD012857.pub2. PMID 35201607
- [Derived] Buitelaar JK, Trott GE, Hofecker M, Waechter S, Berwaerts J, Dejonkheere J, Schauble B. Long-term efficacy and safety outcomes with OROS-MPH in adults with ADHD. Int J Neuropsychopharmacol. 2012 Feb;15(1):1-13. doi: 10.1017/S1461145711001131. Epub 2011 Jul 29. PMID 21798108
- See also: An Open-Label, Multicentre Study to Evaluate the Long-Term Safety of Prolonged Release (PR) OROS Methylphenidate (18, 36, 54, 72 and 90 mg/day) in Adults with Attention Deficit/Hyperactivity Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=47&filename=CR011068_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by Psychiatrists both at medical clinics and private practices between 13-Jan-2006 and 14-Nov-2006
Pre-assignment Details: Subjects who participated in the 42603ATT3002 study and still met all eligibility criteria could enter open-label (OL) phase of this study. Subjects who had received at least 52 weeks of uninterrupted treatment with PR OROS methylphenidate (MPH) and provided informed consent could enter the double-blind phase (DB).45 subjects consented for DB.
Groups:
- Active; Open Label PR OROS MPH: PR OROS MPH 18 to 90 mg once daily
- Placebo: matching placebo
Period: Open Label Phase
Arm/Group | Active | Placebo | Open Label PR OROS MPH
Started | 0 | 0 | 155 (1 screening failure)
Completed | 0 | 0 | 99
Not Completed | 0 | 0 | 56
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 16
Not completed — Withdrawal by Subject | 0 | 0 | 15
Not completed — Lost to Follow-up | 0 | 0 | 11
Not completed — non compliance | 0 | 0 | 5
Not completed — other | 0 | 0 | 6
Period: Double Blind Phase
Arm/Group | Active | Placebo | Open Label PR OROS MPH
Started | 23 | 22 | 0
Completed | 21 | 17 | 0
Not Completed | 2 | 5 | 0
Not completed — Lack of Efficacy | 2 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: Prolonged release (PR) Osmotic Release Oral Systems (OROS) MPH 18 to 90 mg once daily during the OL phase. Subjects who had received at 52 weeks of uninterrupted treatment with PR OROS MPH and provided consent for the DB phase were randomly assigned to placebo or their previous dose of PR OROS MPH (18 to 90 mg once daily)
Arm/Group | Overall Study Population
Number analyzed (Participants) | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 84
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African heritage | 1
  Other: Asian white | 1
  Other: Northern-African + Hindustan | 1
  White | 152
Weight [Mean (Standard Deviation); unit: kg] | 75.1 (16.46)
body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 24.8 (4.47)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: To evaluate the long term safety and tolerability of PR OROS MPH (18, 36, 54, 72 and 90 mg/day) in adults with Attention Deficit Hyperactivity Disorder (ADHD)
Time Frame: Treatment duration for OL extended from 52 wks to 72 wks (International Amendment 2) or 108 wks in Germany. Treatment duration for double-blind (DB) randomized withdrawal: 4 weeks
Population: intent-to-treat: all subjects who used the study medication at least once
Measure: Number; unit: participants
Arm/Group | Active | Placebo | Open Label PR OROS MPH
Number analyzed (Participants) | 23 | 22 | 155
participants
  at least one AE | 7 | 8 | 126
  at least one SAE | 0 | 1 | 12
  at least one severe AE | 0 | 3 | 27
  at least one AE leading to permanent stop | 0 | 0 | 15
  at least one AE leading to temporary stop | 0 | 2 | 23
  at least one AE with concomitant therapy | 0 | 4 | 93
  at least one AE at least possibly related | 3 | 5 | 62

2. Secondary Outcome: Change From OL Baseline to OL Endpoint in Conners' Adult ADHD Rating Scale (CAARS) Total and Subscale Scores
Description: Long term efficacy of PR OROS MPH as assessed by investigator-rated CAARS total score, hyperactivity/impulsivity subscale score and inattention subscale score.
  Subscale scores: best value: 0, worst value: 27
Time Frame: OL baseline, OL endpoint
Population: intent to treat: all subjects who used trial medication at least once
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Placebo | Open Label PR OROS MPH
Number analyzed (Participants) | 0 | 0 | 155
units on a scale
  change from baseline to endpoint in total score |  |  | -1.9 (7.82)
  change from baseline to endpoint in inattention |  |  | -1.0 (4.63)
  change from baseline to endpoint in hyperactivity |  |  | -0.9 (4.36)

3. Primary Outcome: Change From DB Baseline in Conners' Adult ADHD Rating Scale (CAARS) Total Score at DB Endpoint
Description: To evaluate maintenance of treatment effects of PR OROS MPH vs. placebo as measured on CAARS.
  CAARS assesses ADHD symptoms and behaviors in adults. best value: 0 worst value: 54
  Endpoint: last available post-baseline assessment.
Time Frame: DB baseline, DB endpoint
Population: intent to treat: all subjects who used trial medication at least once
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Placebo | Open Label PR OROS MPH
Number analyzed (Participants) | 23 | 22 | 0
units on a scale | 4.0 (7.61) | 6.5 (7.82) |
Statistical Analysis 1: Comparison: Active vs Placebo; Based on preliminary results of a controlled study in adults with MPH, the mean (SD=9) change in CAARS total score from randomization to the 4 week post-randomization endpoint was estimated as +2.5 for PR OROS MPH and +14 for placebo. slightly more conservative, a mean change of 3 in the PR OROS MPH group and a mean increase of 10 in the placebo group were expected. With a two-sided type-I error of 5% and a power of 90%, 37 eligible subjects per group were required; Test type: Superiority or Other; p = 0.2586, ANCOVA — No adjustment for multiplicity was performed. threshold for significance: 0.05 (2-sided); treatment, sex and country as factors, age and baseline sum of inattention and hyperactivity/impulsivity scores as covariate; Mean Difference (Final Values) = 2.89, 95% CI [-2.2055 to 7.9774]

4. Secondary Outcome: Change From OL Baseline in Clinical Global Impression Scale (CGI-S) Score at OL Endpoint
Description: Assessment of the long term effect on overall functioning measured by CGI-S best score: 1 worst score: 7
Time Frame: OL baseline, OL endpoint
Population: intent to treat: all subjects who used trial medication at least once
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Placebo | Open Label PR OROS MPH
Number analyzed (Participants) | 0 | 0 | 155
units on a scale |  |  | -0.3 (1.10)

5. Secondary Outcome: Change From OL Baseline in Quality of Life, Enjoyment and Satisfaction Questionnaire (Q-LES-Q) Score at OL Endpoint
Description: Quality of life measured by Q-LES-Q best score: 100 worst score: 0
Time Frame: OL baseline, OL endpoint
Population: intent to treat: all subjects who used trial medication at least once
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Placebo | Open Label PR OROS MPH
Number analyzed (Participants) | 0 | 0 | 155
units on a scale |  |  | 1.4 (15.15)

6. Secondary Outcome: Change From DB Baseline to DB Endpoint in CGI-S Score
Description: evaluation of treatment effects as rated by the investigator on the CGI-S scale. CGI-S is used to rate the severity of a subject's illness on a 7- point scale ranging from 1 (not ill) to 7 (extremely severe).
Time Frame: DB baseline, DB endpoint
Population: Intent to treat: all subjects who used study medication at least once
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Placebo | Open Label PR OROS MPH
Number analyzed (Participants) | 23 | 22 | 0
units on a scale | 0.6 (1.08) | 1.0 (1.23) |
Statistical Analysis 1: Comparison: Active vs Placebo; Test type: Superiority or Other; p = 0.2616, ANCOVA — No adjustment for multiplicity was performed; ANCOVA on the ranks with sex, treatment and country as factors and age and baseline score as a covariate; Mean Difference (Final Values) = -4.3942, 95% CI [-12.1928 to 3.4044]

7. Secondary Outcome: Change From DB Baseline to DB Endpoint in CAARS Self Rated Scale (CAARS-S:S) Total Score
Description: Evaluation of treatment effects as rated by the subjects on the CAARS-S:S. best score: 0 worst score: 104
Time Frame: DB baseline, DB endpoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Placebo | Open Label PR OROS MPH
Number analyzed (Participants) | 22 | 21 | 0
units on a scale | 4.4 (11.90) | 4.0 (11.98) |
Statistical Analysis 1: Comparison: Active vs Placebo; Test type: Superiority or Other; p = 0.5458, ANCOVA; treatment and country as factors baseline score as covariate; Mean Difference (Final Values) = 2.39, 95% CI [-5.5469 to 10.3213]

ADVERSE EVENTS:
Arm/Group | Active | Placebo | Open Label PR OROS MPH
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/22 | 12/155
Other Adverse Events (participants affected / at risk) | 7/23 | 8/22 | 126/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=23) | Placebo (N=22) | Open Label PR OROS MPH (N=155)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hip surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Lipoma excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Mastectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Whiplash injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Investigation (Investigations) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Breast reconstruction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=23) | Placebo (N=22) | Open Label PR OROS MPH (N=155)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 31 (44)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 10 (12)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 6 (10)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 6 (6)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1) | 12 (14)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 11 (13)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 8 (8)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 7 (9)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (7)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (6)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 33 (54)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 7 (8)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 11 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (7)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (6)
Drug effect decreased (General disorders) | 0 (0) | 0 (0) | 9 (9)
Fatigue (General disorders) | 0 (0) | 1 (1) | 7 (8)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 5 (5)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 4 (5)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 4 (5)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Weight increased (Investigations) | 0 (0) | 1 (1) | 4 (5)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (6)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 6 (6)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 9 (9)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (8)
Impatience (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Impulsive behavior (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Listless (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (2) | 0 (0) | 3 (4)
Stereotypy (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (2) | 1 (1) | 3 (4)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Reticulocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Eyelid edema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Breast reconstruction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Planned sample size for DB phase was 80 subjects. Of 99 subjects at the end of OL phase only 45 subjects consented. No cutoffs for key efficacy assessments in DB entry criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days